CLINICAL TRIAL: NCT03422770
Title: Ultrasonic Markers for Myocardial Fibrosis and Prognosis in Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017/1068
Record Dates: First submitted 2018-01-18; First posted 2018-02-06 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Aortic Valve Stenosis; Myocardial Fibrosis
Keywords: Myocardium; Predictive Value of Tests; Prognosis; Clinical Decision-making; Heart Ventricles; Echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography; Magnetic Resonance Imaging; Hematologic Tests; Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: All participants will undergo 'echo', bloodtests and MRI. Participating patients will in addition undergo electrocardiogram (ECG/Holter ECG) and 6 min walking test.
Who Masked: Outcomes Assessor
Masking Description: Analysis will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild aortic stenosis (Other): 25 patients, all undergoing echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG. All undergoing 1 year control.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test; Diagnostic Test: ECG and Holter-ECG; Diagnostic Test: 6 min walking test
- Moderate aortic stenosis (Other): 25 patients, all undergoing echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG. All undergoing 1 year control.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test; Diagnostic Test: ECG and Holter-ECG; Diagnostic Test: 6 min walking test
- Severe aortic stenosis (Other): 50 patients, all undergoing echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG. All undergoing 1 year control.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test; Diagnostic Test: ECG and Holter-ECG; Diagnostic Test: 6 min walking test
- Controls (Other): 31 subjects, all undergoing echocardiography and blood test and MRI.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Echocardiography — Conventional transthoracic echocardiography will be performed, in addition 3D-imaging and acquisitions with high frame rate. The data from these patients will be anonymized and transferred for post-hoc analysis in dedicated computer software (GE Vingmed, EchoPac 2.0) and in validated machine learning algorithms.
  Other Names: GE Vingmed ultrasound scanner e95, 2017
Diagnostic Test: MRI — Cardiac MRI will be performed. In all patients without contraindications a gadolinium-based contrast agent will be given.
  Other Names: Magnetic resonance imaging
Diagnostic Test: Blood test — Conventional brachial venous blood samples will be drawn. Blood samples will be analyzed for markers of myocardial fibrosis at Oslo University Hospital.The findings will be related to imaging findings.
Diagnostic Test: ECG and Holter-ECG — ECG/Holter-ECG will be performed, and the findings will be related to the imaging findings.
  Arms: Mild aortic stenosis; Moderate aortic stenosis; Severe aortic stenosis
Diagnostic Test: 6 min walking test — 6 MWT will be performed, and the findings will be related to findings from MRI/echocardiography.
  Arms: Mild aortic stenosis; Moderate aortic stenosis; Severe aortic stenosis

SUMMARY:
This study is part of a research project in which new ultrasound-based techniques will be examined to improve clinical decision making for patients with aortic stenosis. These patients could develop increased amounts of myocardial fibrosis. This fibrosis is associated with the patients' prognosis. Fibrosis can be evaluated with magnetic resonance imaging (MRI), which unfortunately is quite expensive and not easily available. Ultrasound-based parameters will be developed for the assessment of the amounts of myocardial fibrosis, especially in the left ventricle. Then it will be examined whether these parameters can predict the patients magnitude of fibrosis and check for association with the patients prognosis. MRI will serve as a gold standard for quantification of myocardial fibrosis. The new echocardiographic techniques and parameters are expected to provide new insights in the interplay between aortic stenosis and left ventricular function, and to ultimately improve the care for patients with aortic stenosis.

The present study's objectives are:

* Quantify the level of myocardial fibrosis in mild, moderate, and severe aortic stenosis compared with a healthy population.
* Evaluate the patients outcome after one and three year of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Able to undergo protocolled investigations
* Patients: Mild, moderate or severe AS

Exclusion Criteria:

* Renal insufficiency
* Previously myocardial infarction (ECG, echocardiogram or hospital record)
* Severe valvular heart disease (except patients)
* Other cardiac disease known to cause myocardial fibrosis
* Severe hypertension
* Other medical conditions deterring protocolled investigation and follow-up
* Other medical conditions affecting 5-yrs prognosis (cancer, pulmonary disease)
* Severely reduced image-quality (echocardiography and MRI)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular morbidity and mortality | 1 + 3 year
  Admission with heart failure or death caused by cardiac disease ('major adverse cardiac events' MACE)

SECONDARY OUTCOMES:
All cause mortality | 3 years
  Mortality in general
Time of first re-hospitalisation | 3 years
  Time of first re-hospitalisation after inclusion
Cardiac systolic function | 1 year.
  Echocardiographic systolic function based on left ventricular ejection fraction, global longitudinal strain, mitral annular plane systolic excursion (MAPSE)
Cardiac diastolic function | 1 year.
  Echocardiographic diastolic function based on the volume of the left atrium, the tricuspidal regurgitation, mitral annular velocities and mitral flow

CONTACTS AND LOCATIONS:
Overall Officials: Svend Aakhus, MD PhD, Study Director — Norwegian University of Science and Technology; Brage Høyem Amundsen, MD PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espeland T, Wigen MS, Dalen H, Berg EAR, Hammer TA, Salles S, Lovstakken L, Amundsen BH, Aakhus S. Mechanical Wave Velocities in Left Ventricular Walls in Healthy Subjects and Patients With Aortic Stenosis. JACC Cardiovasc Imaging. 2024 Feb;17(2):111-124. doi: 10.1016/j.jcmg.2023.07.009. Epub 2023 Sep 6. PMID 37676209
- [Derived] Salles S, Espeland T, Molares A, Aase SA, Hammer TA, Stoylen A, Aakhus S, Lovstakken L, Torp H. 3D Myocardial Mechanical Wave Measurements: Toward In Vivo 3D Myocardial Elasticity Mapping. JACC Cardiovasc Imaging. 2021 Aug;14(8):1495-1505. doi: 10.1016/j.jcmg.2020.05.037. Epub 2020 Aug 26. PMID 32861651